CLINICAL TRIAL: NCT06516549
Title: Impact of Skipping Rope and Informational Pamphlet on Physical Activity Among Adolescents in South Africa
Brief Title: Evaluation of Skipping Rope and Informational Pamphlet Among Adolescents in South Africa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Africa Academy for Public Health (Other); Heidelberg University (Other); Technical University of Munich (Other); USINGA Health and Demographic Surveillance System (Unknown)
Responsible Party: Principal Investigator, Jabulani Ncayiyana, Senior Lecturer/Epidemiologist, University of KwaZulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BREC000064592023
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Moderate-vigorous Physical Activity (MVPA)
Keywords: Physical activity; Skipping rope; Informational pamphlet; Young adolescents; Community; South Africa
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The analyst, or outcome assessor, will be masked in this clinical trial and will not know allocation status until analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Skipping rope and informational pamphlet (Experimental): The intervention group will be provided with a skipping rope and pamphlet with information on the importance of physical activity and ways to engage in physical activity. Both the skipping rope and pamphlet will be provided only once after completing the baseline interview.
  Interventions: Other: Skipping rope and informational pamphlet
- Control (No Intervention): The control arm will not receive provision of intervention (no skipping rope or informational pamphlet).

INTERVENTIONS:
Other: Skipping rope and informational pamphlet — The provision of a skipping rope and an informational pamphlet to the intervention arm participants will happen during the participant interview within the overall DASH cohort study. The enumerator conducting the survey interview will provide each participant in the intervention group with a skipping rope and pamphlet and will read a short script explaining how to use the rope, outlining the main benefits of physical activity for adolescents, and asking participants to read the pamphlet in their own time.
  Arms: Skipping rope and informational pamphlet

SUMMARY:
The purpose of the study is to evaluate the impact of providing a skipping rope and informational pamphlet to adolescents aged 10-14 years on their physical activity intentions and behaviors from baseline to 12-month follow-up when compared with adolescents of the same age who are not provided with any intervention. This study comprises a two-arm randomized controlled trial nested within an adolescent cohort, i.e. a 'randomized trial-within-cohort'. The intervention will include providing each participant with a skipping rope and a pamphlet with general instructions for skipping the rope and messages about the importance of physical activity. The investigators hypothesize that adolescents in a South African community who are provided with a skipping rope and an informational pamphlet on physical activity will engage in more physical activity behaviors and will report greater intentions to be physically active at a 12-month follow-up, compared to a control group of adolescents who do not receive the intervention.

DETAILED DESCRIPTION:
Adolescence is a key period of life during which important physical and psychosocial changes happen. With adolescents comprising about 16% of the world population and 23% of the population in Sub-Saharan Africa (SSA), it is critical to address their health needs to ensure their present wellbeing, as well as healthier trajectories across the life course. One of the most important aspects of a healthy lifestyle during adolescence is physical activity. Regular physical activity improves several physical and mental health outcomes among adolescents. This includes improving muscular strength and flexibility, bone mass, cardiovascular health, lung function, and reducing the risk of obesity and related diseases, such as type 2 diabetes or heart diseases. Additionally, physical activity can improve energy levels, mood, sleep, academic attainment, and social behavior, and it provides an opportunity to connect with peers, by reducing feelings of isolation and fostering friendships.

The World Health Organization (WHO) recommends that adolescents do at least 60 minutes of moderate-to-vigorous physical activity (MVPA) per day, incorporating vigorous-intensity aerobic activities at least three days a week, and limiting the amount of time spent being sedentary. Despite this, research found that adolescents in SSA tend to be largely inactive, with about 82-90% of adolescents reporting low physical activity levels. Similarly, studies suggest that a large proportion of adolescents in South Africa does not meet the physical activity recommendations, with about 93% of males and 95% of females reporting a decrease in physical activity outside of school or sports clubs over adolescence, compared to childhood, and with only 50% of children and adolescents meeting the recommended one hour of MVPA per day.

Skipping, or jumping rope, is a type of physical activity practiced among adolescents across the world. It requires a simple rope and involves the simultaneous rotation of arms and vertical jumping. Skipping rope is an ideal way to promote physical activity among adolescents in South Africa, as it is an easy-to-implement, whole body exercise that has been associated with increased cardiorespiratory fitness and improved bone density. Providing education on the importance of physical activity and instructions on how to skip rope, in addition to the rope itself, can help increase awareness about the benefits of being active and skipping rope, and can help adolescents develop physical activity skills. While there is substantial evidence for short-term positive effects of skipping rope and of successful implementation in schools, there is limited evidence on long-term effects and on implementation in community settings outside of school. Additionally, to the investigators' knowledge, there is limited evidence on skipping rope interventions for adolescents in South Africa.

To address these gaps, the investigators propose to implement a parallel arm randomized controlled trial (1:1 allocation) to promote physical activity among adolescents aged 10-14 years in a community setting in South Africa. This trial will focus on the provision of a skipping rope and informational pamphlet on physical activity and examine their impact on measures of physical activity intentions and behaviors among adolescents over 12 months from baseline. The trial, described in this protocol, will be nested within the Design and Evaluation of Adolescent Health Interventions and Policies (DASH) project, aimed at boosting adolescent health in the SSA region through rigorous population-based intervention and policy research. The DASH project involves the establishment of a cohort of adolescents and young adults, who will be followed up over four waves of data collection in four years. The trial is not invasive.

For the intervention group, the provision of rope and informational pamphlet will happen during the participant interview within the overall DASH cohort study. The fieldworker conducting the survey interview will provide each participant in the intervention group with a rope and pamphlet and will read a short script explaining how to use the rope, outlining the benefits of physical activity for adolescents, and asking participants to read the pamphlet in their own time. The control group will not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Study participant is between ages 10 and 14 years;
* Minors (i.e. less than 18 years of age): the parents or guardians provide written informed consent;
* Minors: the minor participant provides informed assent;
* Study participant is a resident of the study area and intends to stay in the study area for the duration of the study;

Exclusion Criteria:

* Participants with physical disabilities that prevent them from doing physical activity will be excluded;
* Those participants whose capacity to make meaningful decisions is in question because they are "cognitively impaired" will be excluded;
* Individuals with communication difficulties will be excluded.
* Study participants who report suicidal behaviors during baseline data collection will be excluded.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Duration of moderate to vigorous physical activity (MVPA) per week | Baseline and follow up at 12 months after baseline
  Total minutes of MVPA/week. This will be calculated by multiplying the minutes of MVPA on the most recent day participant did MVPA by the number of days MVPA was done.

SECONDARY OUTCOMES:
Proportion of adolescents who meet the MVPA recommendations over the 7 days preceding the interview | Baseline and follow up at 12 months after baseline
  Percentage of adolescents who meet the WHO MVPA recommendations of at least 60 minutes/day of MVPA across the week (>=420 minutes/week)
Intention to engage in physical activity compared to the 7 days preceding the interview | Baseline and follow up at 12 months after baseline
  Intention to engage in physical activity compared to previous 7 days. This will be evaluated by asking participants if they intend to change the amount of physical activity they do in the 7 days following the interview, compared to the 7 days preceding the interview.

OTHER OUTCOMES:
Utilization of rope, process outcome | At the 12-month follow up assessment after baseline
  Utilization modality of skipping rope, that is alone or with friends, among intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Jabulani Ncayiyana, Ph.D., Principal Investigator — University of KwaZulu; Mosa Moshabela, Principal Investigator — University of KwaZulu; Mary Mwanyika-Sando, Principal Investigator — Africa Academy of Public Health; Michael Laxi, Principal Investigator — Technical University of Munich; Till Bärnighausen, Principal Investigator — Heidelberg University; Jacob Burns, Principal Investigator — Technical University of Munich
Locations (1):
- University of KwaZulu-Natal, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available. There are ethical concerns about data privacy and confidentiality that require careful consideration before sharing individual-level data as the trial is embedded with the large DASH Project.
  A detailed statistical plan will be developed in due course and made available on this registry.